CLINICAL TRIAL: NCT05883930
Title: The Effect of Mobile Software "Let's Move" Program Developed Based on Transtheoretical Model on Sedentary Life Behaviors of University Students
Brief Title: The Effect of the Mobile Software Let's Move Program on Changing Sedentary Behaviors of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marmara University (Other)
Collaborators: Marmara University Scientific Research Projects Unit (Unknown); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MARMARA ÜNİVERSİTESİ
Record Dates: First submitted 2023-03-29; First posted 2023-06-01 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Public Health Nursing
Keywords: Physical activity; Mobile software; University students; Public health nursing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transtheoretical Model (TTM)-based "Let's Move" mobile software program (Experimental): Transtheoretical Model (TTM)-based "Let's Move" mobile software program developed for the experimental group will be applied for 12 weeks. Students will be given smart wristbands. Smart wristband data (step numbers) will be integrated into the program. Through this program, students will fill in the pre-test, post-test and follow-up test (at 6 months) and the sedentary lifestyle TTM Sedentary Life Scales (Stages of Change questionnaire, Self-Efficacy and Decision Making scales) and daily step count values.The body mass index, fat and muscle ratios of the students will be evaluated by the researcher. They will be asked to add these values to the program.
  Interventions: Other: 'Let's Move' program
- control group (Experimental): No intervention will be made in the control group. A smart bracelet will be given as a gift in order to follow the step counts of the students. Students will fill in pre-test, post-test and follow-up test (at 6 months) and sedentary lifestyle TTM Sedentary Life Scales (Stages of Change questionnaire, Self-Efficacy and Decision Making scales) and daily step count values via online forms. The body mass index, fat and muscle ratios of the students will be evaluated by the researcher. These values will be recorded.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: 'Let's Move' program — Students will complete data collection forms as part of the program. According to International Physical Activity Questionnaire (IPAQ), those who are low in activity and inactive will be assigned to the appropriate intervention program based on their sedentary lifestyle stage.
  Students will enter the module system prepared according to the five different stages of change [not thinking (1), thinking (2), preparing (3), acting (4), continuing (5)] of sedentary living.
  There are 12 different initiatives for each phase/module of the program. Summary and reinforcing questions are asked at the end of each trial. If participants do not answer the questions, they cannot continue with the next week's initiative.
  Participants' daily step counts with the smart wristband are recorded in the program.
  Daily alerts/reinforcement messages related to that week's initiative will be sent during all phases.
  Other Names: mobile software 'Let's Move' program
  Arms: Transtheoretical Model (TTM)-based "Let's Move" mobile software program
Other: no intervention — No intervention will be applied to the control group.
  Arms: control group

SUMMARY:
Sedentary life means a physically inactive, sedentary life and is the fourth largest risk factor for death worldwide. It is reported that 70% to 85% of young people between the ages of age, representing 15.6% of the population of our country's population, are sedentary. The Transtheoretical Model(TTM) is an easy-to-use and proven model for changing sedentary life. Therefore, in the first stage of this two-stage research, it was aimed to develop the TTM-based 'Let's Move' mobile software program and to test the effect of the mobile software program developed in the second stage on changing the sedentary life behaviors of university students. The universe of this research will consist of 290 students studying at a foundation university in Istanbul. The sample was calculated using the G-power program (3.1.9.4) program. By taking 10% more of the sample, 97 students in the experimental group and 97 students in the control group will be randomly assigned through the Statistical Package for the Social Sciences (SPSS) program. The TTM-based mobile software program "Let's Move" mobile software program developed for the experimental group will be applied for 12 weeks. The effectiveness of the program will be evaluated with the pre-test, post-test and follow-up test, the International Physical Activity Questionnaire, the number of daily steps, the smart bracelet, and the TTM sedentary lifestyle TTM Sedentary Life Scales (Stages of Change, Self-Efficacy and Decision-Making scales). At the end of the research, the effectiveness of the 'Lets's Move' mobile software program "Let's Move" developed in this research in changing the sedentary life will be tested. In addition, it is aimed to increase the number of steps, decrease in sedentary behaviors and make an active lifestyle permanent. All initiatives developed for the TTM sedentary life behavior change stages will be made into a book and the results of the experimental research will be published, contributing and providing evidence to the international literature.

DETAILED DESCRIPTION:
Sedentary lifestyle is an important behavioral problem that threatens health and is reported to be common among young people. University years of study include adolescence and young adulthood. In order to reach the healthy adults of the future, it is very important to spend these periods active, to gain healthy lifestyle behaviors and to make them permanent. Adopting an inactive lifestyle of young people causes many non-communicable diseases (diabetes, hypertension, hyperlipidemia, etc.) later in later ages. For this reason, developing an active lifestyle and changing an inactive lifestyle during the adolescent years are the most important components of reaching healthy societies.

When examining the studies are examined, it is seen that the majority of the studies conducted to reduce sedentary life focus on adults aged > 30 years and a limited number of experimental studies based on the Transtheoretical Model (TTM) for university students.

The Transtheoretical Model argues that change is a process, and not a result, that the individual changes behavior by going through certain stages, and that in order to be successful in change, appropriate initiatives should be planned for the stage of change that the individual is in. The model recommends appropriate biopsychosocial and behavioral interventions by evaluating the individual's readiness for change with the stages of change questionnaire and the self-efficacy and determination levels with scales. It constantly monitors the stage of change that the individual has reached as a result of the initiatives, and offers initiatives to prevent returns and to make the behavior permanent.

ELIGIBILITY:
Inclusion criteria for the study;

* First year students studying in Istanbul Beykent University Vocational School health program between September 2022 and September 2024,
* 18-25 years old,
* Being in the inactive (category 1) and minimally active (category 2) categories according to the International Physical Activity Evaluation Questionnaire,
* Not included in any physical activity program,
* Do not have any physical (orthopedic, chronic diseases, etc.) and mental problems diagnosed by a doctor,
* Accepting the measurement of body weight, height, body fat and muscle ratio and calculation of Body Mass Index (BM) before starting the research, at the 12th week and at the 6th month after its completion,
* Agreeing to use pedometer (pedometer),
* Having an iPhone Operating System (iOs) and android based smart phone,
* Have an active internet connection on their phone,
* Students who voluntarily agree to participate in the research will be formed. Exclusion and Exclusion Criteria;
* Willingness to leave the research.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Baseline
  Physical activity categories by total score Metabolic Equivalent (MET) by IPAQ;
  * Inactive level; 599 MET and below
  * Minimal level; between 600 MET -3000 MET
  * Very active level; 3001 MET and above.
Transtheoretical Model Sedentary Life Stages of Change Survey | Baseline
  Sedentary life change stages constitute the core structure of the Transtheoretical Model. It reflects the individual's attitudes, intentions and behaviors during the change phase. Behavior change; It is a situation assessment consisting of five options and two questions: precontemplation, contemplation, preparation, action and maintenance.
  1. Precontemplation (PC); The individual is either unaware of the problem or has little awareness of it. He has no intention of changing his problematic behavior within 6 months.
  2. Contemplation (C); The individual considers the positive and negative aspects of his/her problematic behavior and is the stage where he/she thinks to change within 6 months.
  3. Preparation (P); The individual intends to change their problematic behavior within 30 days.
  4. Action (A); The individual changed his problematic behaviors within 6 months.
  5. Maintenance (M); The individual has changed his unhealthy behavior 6 months ago at this stage.
Transtheoretical Model Sedentary Life Self-efficacy Scale | Baseline
  Self-efficacy Scale; It is an individual's belief about himself/herself that he/she can successfully perform a certain behavior, and it reflects self-confidence. The scale consists of 6 items that include self-confidence in quitting sedentary behavior. It is a five-point Likert type. It ranges from 1: Not at all trusting to 5: Very confident. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on the self-efficacy scale indicates that the student's self-efficacy in changing sedentary life behavior has increased.
Transtheoretical Model Sedentary Life Decision Balance Scale | Baseline
  The decision-making scale consists of two sub-dimensions that measure the benefits and harms of making a behavior change decision.
  * Sedentary life behavior change decision-making benefit perception sub-dimension; It consists of 1, 3, 5, 7, 9, and 11 items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that they are aware of the benefits of behavior change and that they are more likely to change their behavior.
  * Sedentary life behavior change decision making harm sub-dimension; It consists of the 2nd, 4th, 6th, 8th, 10th, and 12th items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that the harms of behavior change attract more attention and the probability of changing behavior is less.
Step counter | Baseline
  Categories of steps per day Number of steps per day-Category less than 2500 steps-"basal activity" 2500-4999 steps- "limited activity" Those taking 5000-7499 steps- "little activity" 7500-9999 steps-"somewhat active" 10000-12499 steps taken- "active" Those who take more than 12500 steps- "highly active"
Body Mass Index (BMI) | Baseline
  According to the World Health Organization's body mass index data, individuals below 18.5 kg/m2 are considered "thin," values between 18.5and 24.99 are considered "normal," 25.0to 29.9 kg/m2 are considered "mildly obese," and 30.0 kg/m2 or more are considered "obese." After completion of the study, participants will be evaluated according to their body mass index.
Body fat to muscle ratio | Baseline
  For men and women to be physically and psychosocially healthy, the ratio of standard oils (essential oils) should be 15% for men and 23% for women.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 12th weekend
  Physical activity categories by total score Metabolic Equivalent (MET) by IPAQ;
  * Inactive level; 599 MET and below
  * Minimal level; between 600 MET -3000 MET
  * Very active level; 3001 MET and above.
Transtheoretical Model Sedentary Life Stages of Change Survey | 12th weekend
  Sedentary life change stages constitute the core structure of the Transtheoretical Model. It reflects the individual's attitudes, intentions and behaviors during the change phase. Behavior change; It is a situation assessment consisting of five options and two questions: precontemplation, contemplation, preparation, action and maintenance.
  1. Precontemplation (PC); The individual is either unaware of the problem or has little awareness of it. He has no intention of changing his problematic behavior within 6 months.
  2. Contemplation (C); The individual considers the positive and negative aspects of his/her problematic behavior and is the stage where he/she thinks to change within 6 months.
  3. Preparation (P); The individual intends to change their problematic behavior within 30 days.
  4. Action (A); The individual changed his problematic behaviors within 6 months.
  5. Maintenance (M); The individual has changed his unhealthy behavior 6 months ago at this stage.
Transtheoretical Model Sedentary Life Self-efficacy Scale | 12th weekend
  It is an individual's belief about himself/herself that he/she can successfully perform a certain behavior, and it reflects self-confidence. The scale consists of 6 items that include self-confidence in quitting sedentary behavior. It is a five-point Likert type. It ranges from 1: Not at all trusting to 5: Very confident. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on the self-efficacy scale indicates that the student's self-efficacy in changing sedentary life behavior has increased.
Transtheoretical Model Sedentary Life Decision Balance Scale | 12th weekend
  The decision-making scale consists of two sub-dimensions that measure the benefits and harms of making a behavior change decision.
  * Sedentary life behavior change decision-making benefit perception sub-dimension; It consists of 1, 3, 5, 7, 9, and 11 items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that they are aware of the benefits of behavior change and that they are more likely to change their behavior.
  * Sedentary life behavior change decision making harm sub-dimension; It consists of the 2nd, 4th, 6th, 8th, 10th, and 12th items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that the harms of behavior change attract more attention and the probability of changing behavior is less.
Step counter | 12th weekend
  Categories of steps per day Number of steps per day-Category less than 2500 steps-"basal activity" 2500-4999 steps- "limited activity" Those taking 5000-7499 steps- "little activity" 7500-9999 steps-"somewhat active" 10000-12499 steps taken- "active" Those who take more than 12500 steps- "highly active"
Body Mass Index (BMI) | 12th weekend
  According to the World Health Organization's body mass index data, individuals below 18.5 kg/m2 are considered "thin," values between 18.5and 24.99 are considered "normal," 25.0to 29.9 kg/m2 are considered "mildly obese," and 30.0 kg/m2 or more are considered "obese." After completion of the study, participants will be evaluated according to their body mass index.
Body fat to muscle ratio | 12th weekend
  For men and women to be physically and psychosocially healthy, the ratio of standard oils (essential oils) should be 15% for men and 23% for women.

OTHER OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 24th weekend.
  Physical activity categories by total score Metabolic Equivalent (MET) by IPAQ;
  * Inactive level; 599 MET and below
  * Minimal level; between 600 MET -3000 MET
  * Very active level; 3001 MET and above.
Transtheoretical Model Sedentary Life Stages of Change Survey | 24th weekend.
  Sedentary life change stages constitute the core structure of the Transtheoretical Model. It reflects the individual's attitudes, intentions and behaviors during the change phase. Behavior change; It is a situation assessment consisting of five options and two questions: precontemplation, contemplation, preparation, action and maintenance.
  1. Precontemplation (PC); The individual is either unaware of the problem or has little awareness of it. He has no intention of changing his problematic behavior within 6 months.
  2. Contemplation (C); The individual considers the positive and negative aspects of his/her problematic behavior and is the stage where he/she thinks to change within 6 months.
  3. Preparation (P); The individual intends to change their problematic behavior within 30 days.
  4. Action (A); The individual changed his problematic behaviors within 6 months.
  5. Maintenance (M); The individual has changed his unhealthy behavior 6 months ago at this stage.
Transtheoretical Model Sedentary Life Self-efficacy Scale | 24th weekend.
  It is an individual's belief about himself/herself that he/she can successfully perform a certain behavior, and it reflects self-confidence. The scale consists of 6 items that include self-confidence in quitting sedentary behavior. It is a five-point Likert type. It ranges from 1: Not at all trusting to 5: Very confident. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on the self-efficacy scale indicates that the student's self-efficacy in changing sedentary life behavior has increased.
Transtheoretical Model Sedentary Life Decision Balance Scale | 24th weekend.
  The decision-making scale consists of two sub-dimensions that measure the benefits and harms of making a behavior change decision.
  * Sedentary life behavior change decision-making benefit perception sub-dimension; It consists of 1, 3, 5, 7, 9, and 11 items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that they are aware of the benefits of behavior change and that they are more likely to change their behavior.
  * Sedentary life behavior change decision making harm sub-dimension; It consists of the 2nd, 4th, 6th, 8th, 10th, and 12th items of the scale. The minimum score to be taken from these scales will be '6' and the maximum score will be '30'. A high score on this sub-dimension indicates that the harms of behavior change attract more attention and the probability of changing behavior is less.
Step counter | 24th weekend.
  Categories of steps per day Number of steps per day-Category less than 2500 steps-"basal activity" 2500-4999 steps- "limited activity" Those taking 5000-7499 steps- "little activity" 7500-9999 steps-"somewhat active" 10000-12499 steps taken- "active" Those who take more than 12500 steps- "highly active"
Body Mass Index (BMI) | 24th weekend
  According to the World Health Organization's body mass index data, individuals below 18.5 kg/m2 are considered "thin," values between 18.5and 24.99 are considered "normal," 25.0to 29.9 kg/m2 are considered "mildly obese," and 30.0 kg/m2 or more are considered "obese." After completion of the study, participants will be evaluated according to their body mass index.
Body fat to muscle ratio | 24th weekend
  For men and women to be physically and psychosocially healthy, the ratio of standard oils (essential oils) should be 15% for men and 23% for women.

CONTACTS AND LOCATIONS:
Overall Officials: GÖZDE ÖZDEMİR, Principal Investigator — https://www.marmara.edu.tr/; SAİME EROL, Study Director — https://www.marmara.edu.tr/
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University/ Maltepe, Maltepe, Istanbul
  - Marmara University/ Maltepe, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
At the end of the 12th week and the 24th week, the results of the research will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 13.06.2023-13.09.2023
Access Criteria: It can be seen on the page where randomized controlled trial (RCT) data are shared.
URL: https://clinicaltrials.gov/

REFERENCES:
- [Result] Han H, Gabriel KP, Kohl HW. Evaluations of Validity and Reliability of a Transtheoretical Model for Sedentary Behavior among College Students. Am J Health Behav. 2015 Sep;39(5):601-9. doi: 10.5993/AJHB.39.5.2. PMID 26248170
- [Result] Kim H, Kohl Iii HW, Pettee Gabriel KK, Han H. Differential Use of Strategic Constructs of the Transtheoretical Model across Accelerometer-determined Sedentary Time. Am J Health Behav. 2020 Jan 1;44(1):18-25. doi: 10.5993/AJHB.44.1.3. PMID 31783929
- [Result] Lee JS, Kang MA, Lee SK. Effects of the e-Motivate4Change Program on Metabolic Syndrome in Young Adults Using Health Apps and Wearable Devices: Quasi-Experimental Study. J Med Internet Res. 2020 Jul 30;22(7):e17031. doi: 10.2196/17031. PMID 32729838
- [Result] Kleis RR, Hoch MC, Hogg-Graham R, Hoch JM. The Effectiveness of the Transtheoretical Model to Improve Physical Activity in Healthy Adults: A Systematic Review. J Phys Act Health. 2021 Jan 1;18(1):94-108. doi: 10.1123/jpah.2020-0334. Epub 2020 Dec 1. PMID 33260143
- [Result] Chen P, Mao L, Nassis GP, Harmer P, Ainsworth BE, Li F. Coronavirus disease (COVID-19): The need to maintain regular physical activity while taking precautions. J Sport Health Sci. 2020 Mar;9(2):103-104. doi: 10.1016/j.jshs.2020.02.001. Epub 2020 Feb 4. No abstract available. PMID 32099716
- [Result] Wu YK, Chu NF. Introduction of the transtheoretical model and organisational development theory in weight management: A narrative review. Obes Res Clin Pract. 2015 May-Jun;9(3):203-13. doi: 10.1016/j.orcp.2014.12.003. Epub 2015 Jan 5. PMID 25571777
- [Result] Han H, Pettee Gabriel K, Kohl HW 3rd. Application of the transtheoretical model to sedentary behaviors and its association with physical activity status. PLoS One. 2017 Apr 27;12(4):e0176330. doi: 10.1371/journal.pone.0176330. eCollection 2017. PMID 28448531
- [Result] Kim H, Park E, Lee S, Kim M, Park EJ, Hong S. Self-Management of Chronic Diseases Among Older Korean Adults: An mHealth Training, Protocol, and Feasibility Study. JMIR Mhealth Uhealth. 2018 Jun 29;6(6):e147. doi: 10.2196/mhealth.9988. PMID 29959109
- [Result] Wang JB, Cadmus-Bertram LA, Natarajan L, White MM, Madanat H, Nichols JF, Ayala GX, Pierce JP. Wearable Sensor/Device (Fitbit One) and SMS Text-Messaging Prompts to Increase Physical Activity in Overweight and Obese Adults: A Randomized Controlled Trial. Telemed J E Health. 2015 Oct;21(10):782-92. doi: 10.1089/tmj.2014.0176. Epub 2015 Jun 2. PMID 26431257
- [Result] Andersen LB, Harro M, Sardinha LB, Froberg K, Ekelund U, Brage S, Anderssen SA. Physical activity and clustered cardiovascular risk in children: a cross-sectional study (The European Youth Heart Study). Lancet. 2006 Jul 22;368(9532):299-304. doi: 10.1016/S0140-6736(06)69075-2. PMID 16860699
- [Result] Kim BH, Lee H. Associations Between Smartphone Use for Physical Activity by South Korean College Students and Behavioral Change Constructs of the Transtheoretical Model. Percept Mot Skills. 2022 Aug;129(4):1270-1282. doi: 10.1177/00315125221099258. Epub 2022 May 6. PMID 35522152
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Result] Tudor-Locke C, Washington TL, Hart TL. Expected values for steps/day in special populations. Prev Med. 2009 Aug;49(1):3-11. doi: 10.1016/j.ypmed.2009.04.012. Epub 2009 May 4. PMID 19409409
- See also: World Health Organization, 2020, Physical Activity — https://www.who.int/news-room/fact-sheets/detail/physical-activity
- See also: World Health Organization, 2021, Body Mass Index (BMI) — https://www.who.int/data/gho/data/themes/theme-details/gho/body-mass-index-(bmi)
- See also: World Health Organization, 2020, Adolescent And Young Adult Health — https://www.who.int/news-room/fact-sheets/detail/adolescents-health-risks-and-solutions
- Available data/document: Scales Validity and Reliability — https://tr-scales.arabpsychology.com/wp-content/uploads/pdf/uluslararasi-fiziksel-aktivite-anketi-toad.pdf — Ozturk, M. (2005). The validity and reliability of the international physical activity questionnaire and the determination of physical activity level in university students. Unpublished master thesis. Hacettepe University, Institute of Health Sciences, Ankara.

DOCUMENTS (2):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT05883930/Prot_000.pdf
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT05883930/ICF_001.pdf